CLINICAL TRIAL: NCT01431898
Title: A Phase 1b, Randomized, Single-Blind, Multiple-Dose Ranging Study Evaluating the Safety, Tolerability, Pharmacokinetics and Antiviral Activity of GS-9669 in Subjects With Chronic Hepatitis C Virus Infection
Brief Title: Safety, Tolerability, Pharmacokinetics and Antiviral Activity of GS-9669 in Subjects With Chronic Hepatitis C Virus Infection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Masking: Single | Purpose: Treatment
Other Study IDs: GS-US-257-0102
Record Dates: First submitted 2011-09-01; First posted 2011-09-12 (Estimated); Last update posted 2012-07-25 (Estimated); Status verified 2012-03

CONDITIONS: Hepatitis C
Keywords: HCV RNA; Polymerase inhibitor; Treatment naïve and Treatment experienced; GS-9669; Hepatitis C; HCV
MeSH Terms: conditions — Hepatitis C | interventions — GS-9669; Food; Communication Devices for People with Disabilities; WW Domain-Containing Oxidoreductase

STUDY DESIGN:
Who Masked: Participant

ARMS (1):
- Multiple-dose, dose-escalation study of GS-9669 (Experimental): Multiple-dose, dose-escalation study of GS-9669, a nonnucleotide NS5B inhibitor of hepatitis C virus (HCV), in subjects with chronic HCV infection. Dosing is planned in up to 7 unique dosing cohorts. Each cohort will be comprised of 10 genotype 1a (Cohorts 1, 2, 3, 4, and 5) or genotype 1b (Cohort 6 and 7), with eight subjects randomized to receive active drug and two subjects randomized to receive placebo per cohort.
  Interventions: Drug: GS-9669 tablets; Drug: Placebo to Match GS-9669 tablet

INTERVENTIONS:
Drug: GS-9669 tablets
  Other Names: Cohort 1 (N = 10, genotype 1a): 100 mg GS-9669 or placebo BID with; food [total daily dose (TDD) = 200 mg] for 3 days;; Cohort 2 (N = 10, genotype 1a): 400 mg GS-9669 or placebo BID with; food (TDD = 800 mg) for 3 days;; Cohorts 1 and 2 may be conducted in parallel. Additional adaptive BID; and/or QD cohorts (Cohorts 3-5) in genotype 1a subjects may be; conducted depending on the safety, virology, and available; pharmacokinetics from the first two cohorts. Cohorts 3 -5 may be; conducted in parallel if the total daily dose is lower than the highest total; daily dose previously tested and determined to be safe and well tolerated.; Cohort 3 (N = 10, genotype 1a): up to 400 mg GS-9669 or placebo BID; with food (TDD = up to 800 mg) for 3 days;; Cohort 4 (N = 10, genotype 1a): up to 400 mg GS-9669 or placebo BID; Cohort 5 (N=10, genotype 1a): up to 800 mg GS-9669 or placebo QD in; the morning with food (TDD = up to 800 mg) for 3 days;; Based on the results of Cohorts 1 to 5, one or more regimens will be; selected for an evaluation in genotype 1b subjects to enable comparison; between genotypes. Cohorts 6 and 7 may proceed in parallel with other; Cohorts if the total daily dose is the same or lower than the highest total; Cohort 6 (N = 10, genotype 1b): up to 400 mg GS-9669 or placebo BID; with food (TDD = up to 800 mg) for 3 days; Cohort 7 (N = 10, genotype 1b): up to 800 mg GS-9669 or placebo QD in; the morning with food (TDD = up to 800 mg) for 3 days.
Drug: Placebo to Match GS-9669 tablet

SUMMARY:
This is a research study to evaluate the safety, tolerability and anti-viral activity of GS-9669 in patients with Hepatitis C infection.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects 18-65 years of old, inclusive
* Documented chronic HCV infection to be of at least 6 months duration and plasma HCV RNA ≥ 5 log10 IU/mL at screening.
* HCV treatment naïve or PEG-IFN, IFN, and/or RBV experienced (treatment must have ceased at least 3 months prior to screening). Treatment experienced subjects should not exceed 40% of the subjects enrolled in each cohort
* Mono-infection with HCV genotype 1a for Cohorts 1, 2, 3, 4, and 5 and mono-infection with HCV genotype 1b for Cohort 6 and 7.
* Estimated creatinine clearance ≥ 70 mL/min,
* QTcF interval ≤ 450 msec for males and ≤ 470 msec for females, QRS duration < 120 msec, PR interval < 220 msec,
* Body mass index (BMI) of 19.0 to 34.0 kg/m^2, inclusive.

Exclusion Criteria:

* Urine drug screen positive for illicit/illegal drugs
* ALT and AST levels > 5 times the upper limit of the normal range (ULN)
* Direct bilirubin > ULN, clinical or other laboratory evidence of hepatic decompensation (i.e., platelets < 90,000/mm^3, prothrombin time ≥ 1.5 × ULN and albumin < 3.5 g/dL) are not eligible for study participation.
* Subjects with an absolute neutrophil count (ANC) < 1,000 cells/mm^3 (< 750 cells/mm^3 for black or African-American subjects), hemoglobin (Hb) < 11 g/dL,
* Coinfected with hepatitis B virus (HBV), human immunodeficiency virus (HIV), or another HCV genotype other than genotype 1a/b are not eligible for study participation.
* Evidence of hepatocellular carcinoma (e.g., a-fetoprotein > 50 ng/mL or as indicated by recent ultrasound or other standard of care measure)
* History of significant cardiac disease. The following ECG abnormalities at screening are exclusionary: QTcF (QT corrected using Fridericia's formula=QT/RR^0.333) > 450 msec for males and > 470 for females; QRS > 120 msec (left or right hemiblock is not exclusionary); PR interval > 220 msec; bradycardia (< 45 beats per minute); second or third degree heart block.
* History of clinically-significant illness or any other major medical disorder that may interfere with subject treatment, assessment or compliance with the protocol
* History of a primary gastrointestinal disorder that could interfere with the absorption of the study drug or that could interfere with normal gastrointestinal anatomy or motility

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2011-09; Primary Completion 2011-12 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability | through 24 weeks of off-treatment follow-up
  To evaluate safety and tolerability of escalating multiple oral doses of GS 9669.
  Safety will be assessed during the study through the reporting of adverse events, clinical laboratory tests, physical examinations, vital signs, and 12-lead ECGs at various time points during the study.
Antiviral Activity | through 24 weeks of off-treatment follow-up
  To evaluate antiviral activity of GS-9669 against HCV in genotype-1a and 1b (GT1a/b) subjects. This will be evaluated using change from baseline in plasma HCV RNA. Reduction in HCV RNA will be summarized as categorical (as < 1, ≥ 1 to <2, ≥ 2 to <3, or ≥ 3 log10 IU/mL) reduction from baseline.

SECONDARY OUTCOMES:
Viral Dynamics and Pharmacodynamics | Through 17 days of therapy
  To characterize the viral dynamics of GS-9669. The median change from baseline in HCV RNA and time-weighted average change from baseline through Day 3 will be assessed based on plasma HCV RNA sampling times to characterize the viral dynamics of GS-9669.
composite of Pharmacokinetics | Through 17 days of therapy
  To characterize the plasma PK parameters of GS-9669. The secondary PK endpoints will be evaluated using standard non-compartmental methods. Relevant PK parameters will be determined using standard non-compartmental methods with the linear-logarithmic trapezoidal rule utilizing a PK data analysis program (e.g., WinNonlin®) for GS-9669 as appropriate: Cmax, Tmax, Clast, Tlast, Ctau, λz, AUC0-last, AUCtau, , CL/F, and T½.
Genotypic Changes | through 24 weeks of off-treatment follow-up
  To characterize genotypic changes from baseline in the NS5B coding region of HCV following multiple dose administration of GS-9669 and for up to 24 weeks thereafter

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Rossi, PharmD, Study Director — Gilead Sciences
Locations (11):
- United States (10):
  - Impact Clinical Trials, Los Angeles, California
  - Avail Clinical Research, LLC, DeLand, Florida
  - Orlando Clinical Research Center, Orlando, Florida
  - Impact Clinical Trials, Las Vegas, Nevada
  - CRI Worldwide, Willingboro, New Jersey
  - CRI Worldwide, Philadelphia, Pennsylvania
  - Alamo Medical Research, San Antonio, Texas
  - Lifetree Clinical Research, LC, Salt Lake City, Utah
  - University of Utah Health Sciences Center, Salt Lake City, Utah
  - Charles River Clinical Services Northwest, Tacoma, Washington
- Fundacion de Investigacion de Diego, San Juan, Puerto Rico

REFERENCES:
- [Derived] Dvory-Sobol H, Voitenleitner C, Mabery E, Skurnac T, Lawitz EJ, McHutchison J, Svarovskaia ES, Delaney W, Miller MD, Mo H. Clinical and in vitro resistance to GS-9669, a thumb site II nonnucleoside inhibitor of the hepatitis C virus NS5B polymerase. Antimicrob Agents Chemother. 2014 Nov;58(11):6599-606. doi: 10.1128/AAC.02815-14. Epub 2014 Aug 25. PMID 25155588
- [Derived] Fenaux M, Eng S, Leavitt SA, Lee YJ, Mabery EM, Tian Y, Byun D, Canales E, Clarke MO, Doerffler E, Lazerwith SE, Lew W, Liu Q, Mertzman M, Morganelli P, Xu L, Ye H, Zhang J, Matles M, Murray BP, Mwangi J, Zhang J, Hashash A, Krawczyk SH, Bidgood AM, Appleby TC, Watkins WJ. Preclinical characterization of GS-9669, a thumb site II inhibitor of the hepatitis C virus NS5B polymerase. Antimicrob Agents Chemother. 2013 Feb;57(2):804-10. doi: 10.1128/AAC.02052-12. Epub 2012 Nov 26. PMID 23183437